CLINICAL TRIAL: NCT00122538
Title: HAART Regimen Comprising 3TC + ddI + EFV in Once-daily Administration in HIV-1 Infected Children in Burkina Faso
Brief Title: Once-daily Highly Active Antiretroviral Treatment Regimen Administration in HIV-1 Infected Children in Burkina Faso (ANRS 12103 BURKINAME)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12103 BURKINAME
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infections; AIDS
Keywords: HAART; once-daily; child; africa; HIV; AIDS; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — efavirenz; Lamivudine; Didanosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Efavirenz (EFV)
Drug: Lamivudine (3TC)
Drug: Didanosine (ddI)

SUMMARY:
The purpose of this study is to try a known antiretroviral combination in HIV- infected children with only one intake a day, in order to simplify the prescription and improve adherence to treatment. This is what is called a phase II clinical trial, only recruiting and following a small number of children (50) during one year to evaluate the quantity of drug in the blood just before it is taken and one to three hours after it is taken. The other important objective is to study the tolerance of drugs in that mode of prescription of the triple combination.

DETAILED DESCRIPTION:
The data relating to pharmacology tolerance and efficacy of the once-daily combination of 3TC + ddI + EFV have never been studied.

This regimen may lead to a better treatment of the HIV-1 infected children in developing countries, as well as in Europe. Because of its simplicity it would facilitate observance that is one of the essential parameters of efficacy of treatments.

The main objectives are those of a phase II clinical trial:

* Assess the virological and immunological efficacy of a once daily HAART regimen comprising lamivudine (3TC) + didanosine (ddI) + efavirenz (EFV) [pediatric reference];
* Analyse the pharmacological characteristics of this combination in children;
* Assess the tolerance;
* Study the appearance of resistance;
* Evaluate the observance to treatment.

  50 HIV-1 infected children aged 30 months to 15 years whose clinical and immunological state (stage B or C) requires antiretroviral treatment, will be included in the study. They should be naive of any ARV treatment (except the treatment received in the framework of PMTCT (Prevention of Mother to Child Transmission).

Data Collection and Development of the Study:

* Monthly clinical examination;
* RNA HIV-1 and CD4 counts;
* Pharmacological dosages;
* Haematology and biochemistry surveillance;
* Genotypic resistance at inclusion; and, in case of unsuccess or failure,
* Assessment of observance according to alternate methods.

Laboratory examinations will be carried out at Centre Muraz except for genotyping and for pharmacological tests sent to Montpellier Teaching Hospital (France).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected children
* Weight over 12 kgs
* Age over 30 months
* Clinical stage requiring HAART
* Naive to antiretroviral treatment (except PMTCT prophylaxis)
* Mother's or tutor's informed consent signed

Exclusion Criteria:

* HIV-2 or dual HIV infection
* Previous antiretroviral therapy
* Children unable to swallow pills
* Known resistance to non-nucleoside reverse transcriptase inhibitor (NNRTI)

Ages: 30 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with HIV RNA less than 400 copies per ml and less than 50 copies per ml at month 12 (M12) | 12 and 24 months
Cmin and Cmax for the three drugs | 15 days
Grade 3 or 4 undesirable effects frequency | through out the trial

SECONDARY OUTCOMES:
Percentage of patients with CD4 greater than 25 percent at M12 and M24 | 12 and 24 months
Amplitude of viral load reduction | 12 and 24 months
Slope of CD4 compared with the initial values | 12 and 24 months
Percentage of patients lost to follow-up | 12 and 24 months
Percentage of deaths and of B or C classing events | Through out the trial
Percentage of treatment interruption | Through out the trial
Percentage and type of resistance mutations | 12 and 24 months
Percentage of patients forgetting more than one pill within the last three days | Through out the trial

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Msellati, MD, PhD, Study Chair — Institut de Recherche et de Développement (IRD UMR 145); Aboubacar Nacro, MD, Principal Investigator — CHU Sanou Souro, Bobo-Dioulasso
Locations (1):
- Service de pediatrie, CHU Sanou Souro, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Derived] Bouazza N, Treluyer JM, Msellati P, Van de Perre P, Diagbouga S, Nacro B, Hien H, Zoure E, Rouet F, Ouiminga A, Blanche S, Hirt D, Urien S. A novel pharmacokinetic approach to predict virologic failure in HIV-1-infected paediatric patients. AIDS. 2013 Mar 13;27(5):761-8. doi: 10.1097/QAD.0b013e32835caad1. PMID 23719348
- [Derived] Barro M, Some J, Foulongne V, Diasso Y, Zoure E, Hien H, Francois R, Michel S, Drabo A, Tamboura H, Ouiminga A, Diagbouga S, Hien A, Yameogo S, Van De Perre P, Nacro B, Msellati P. Short-term virological efficacy, immune reconstitution, tolerance, and adherence of once-daily dosing of didanosine, lamivudine, and efavirenz in HIV-1-infected African children: ANRS 12103 Burkiname. J Acquir Immune Defic Syndr. 2011 Jul 1;57 Suppl 1:S44-9. doi: 10.1097/QAI.0b013e31821fd64f. PMID 21857286
- [Derived] Bouazza N, Hirt D, Bardin C, Diagbouga S, Nacro B, Hien H, Zoure E, Rouet F, Ouiminga A, Blanche S, Van De Perre P, Treluyer JM, Msellati P, Urien S. Is the recommended once-daily dose of lamivudine optimal in West African HIV-infected children? Antimicrob Agents Chemother. 2010 Aug;54(8):3280-6. doi: 10.1128/AAC.00306-10. Epub 2010 Jun 1. PMID 20516271